CLINICAL TRIAL: NCT02146053
Title: Validation of a Simple Questionnaire to Assess Gastrointestinal Symptoms After Oral Ferrous Sulphate Supplementation.
Brief Title: Questionnaire to Assess Gastrointestinal Symptoms of Oral Iron.
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Medical Research Council (Other Government)
Collaborators: King's College London (Other)
Responsible Party: Principal Investigator, dora pereira, Dr, Medical Research Council
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: Symptoms KCL
Record Dates: First submitted 2014-05-21; First posted 2014-05-23 (Estimated); Last update posted 2017-02-06 (Estimated); Status verified 2017-02

CONDITIONS: Anemia; Constipation; Diarrhea; Abdominal Pain; Heartburn; Side Effect
Keywords: healthy participants; gastrointestinal side-effects associated with oral iron
MeSH Terms: conditions — Anemia; Constipation; Diarrhea; Abdominal Pain; Heartburn | interventions — ferrous sulfate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ferrous sulfate (Active Comparator): ferrous sulfate taken at mealtimes twice daily during 1 week of the treatment period.
  Interventions: Dietary Supplement: ferrous sulfate
- Placebo (Placebo Comparator): placebo taken at mealtimes twice daily during 1 week of the treatment period.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: ferrous sulfate — ferrous sulphate (200 mg capsules containing 65 mg of iron) to be taken at mealtimes twice daily for 7 days during the treatment period.
  Other Names: ferrous sulphate
  Arms: Ferrous sulfate
Dietary Supplement: Placebo — placebo capsules: methyl cellulose
  Arms: Placebo

SUMMARY:
Oral iron supplementation is often associated with rapid onset of gastrointestinal side-effects. The aim of this study was to develop and trial a short, simple questionnaire to capture these early side-effects and to determine which symptoms are more discriminating.

The study was a double-blind placebo-controlled randomized parallel trial with one week treatment followed by one week wash-out. Subjects were randomized into two treatment groups (n=10/group) to receive either ferrous sulphate (200 mg capsules containing 65 mg of iron) or placebo, both to be taken at mealtimes twice daily during the treatment period. Subjects completed the questionnaires daily for 14 days. The questionnaire included gastrointestinal symptoms commonly reported to be associated with the oral intake of ferrous iron salts (i.e. nausea, vomiting, heartburn, abdominal pain, diarrhoea, and constipation).

ELIGIBILITY:
Inclusion Criteria:

* Generally healthy subjects.

Exclusion Criteria:

* The presence of any chronic disease, pregnancy or lactation were considered as exclusion criteria.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2004-03; Primary Completion 2004-12 (Actual); Study Completion 2004-12 (Actual)

PRIMARY OUTCOMES:
gastrointestinal symptoms | 14 days
  Subjects completed the questionnaires daily for 14 days. The questionnaire included gastrointestinal symptoms commonly reported to be associated with the oral intake of ferrous iron salts (i.e. nausea, vomiting, heartburn, abdominal pain, diarrhoea, and constipation).

CONTACTS AND LOCATIONS:
Overall Officials: Miranda Lomer, PhD, Principal Investigator — King's College London; Jonathan Powell, PhD, Study Chair — MRC Human Nutrition Research
Locations (1):
- King's College London, London, United Kingdom

REFERENCES:
- [Derived] Pereira DI, Couto Irving SS, Lomer MC, Powell JJ. A rapid, simple questionnaire to assess gastrointestinal symptoms after oral ferrous sulphate supplementation. BMC Gastroenterol. 2014 Jun 4;14:103. doi: 10.1186/1471-230X-14-103. PMID 24899360